CLINICAL TRIAL: NCT01490944
Title: Impact of Vitamin B12 Supplementation With Iron and Folic Acid on Adolescent Girls
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indian Council of Medical Research (Other Government)
Collaborators: Delhi University (Other)
Responsible Party: Principal Investigator, G.S.Toteja, Scientist-F (Deputy Director General, Senior Grade) and Principal Investigator, Indian Council of Medical Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNRT/Ph.D/4/2010; 3/1/2/34/10-RHN (Other Grant/Funding Number: Indian Council of Medical Research)
Record Dates: First submitted 2011-12-11; First posted 2011-12-13 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-01

CONDITIONS: Anaemia
MeSH Terms: conditions — Anemia | interventions — Iron; Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron and Folic Acid (Active Comparator)
  Interventions: Drug: Iron and Folic Acid
- Iron, Folic acid and cyanocobalamin (Experimental)
  Interventions: Drug: Iron, Folic acid and Cyanocobalamin

INTERVENTIONS:
Drug: Iron, Folic acid and Cyanocobalamin — Total duration= 6 months Iron=100 mg, Folic acid= 500 mcg, Cyanocobalamin 500 mcg weekly supplementation in the form of capsule for 6 weeks
  Iron=100 mg, Folic acid= 500 mcg, Cyanocobalamin 15 mcg weekly supplementation in the form of capsule for next 20 weeks
  Arms: Iron, Folic acid and cyanocobalamin
Drug: Iron and Folic Acid — Iron= 100 mg, Folic acid= 500 mcg weekly supplementation in the form of capsule for 6 months
  Arms: Iron and Folic Acid

SUMMARY:
The study is a clinical trial to assess the effectiveness of Vitamin B12 supplementation along with Iron Folic Acid (IFA) in combating anaemia. Adolescent anaemic girls will be randomly divided into two groups.

* Group 1: IFA weekly supplementation along with Information, Education, Communication sessions
* Group 2: IFA + Cyanocobalamin weekly supplementation along with Information, Education, Communication sessions

Duration of supplementation: 6 months

DETAILED DESCRIPTION:
The study is a randomized clinical trial to be conducted on mild or moderately anaemic adolescent girls (11-18 yrs) in a slum in Delhi. Anaemic adolescent girls (n=360) will be randomly divided into two groups. Group 1(n=180) will be given weekly supplementation of Iron (100 mg) and Folic acid (500 mcg) for six months, whereas group 2 (n=180) will be given weekly supplementation of Iron Folic Acid and cyanocobalamin (Vitamin B12) to assess the impact of Vitamin B12 supplementation on reducing the prevalence of anaemia. For first six weeks, 500 mcg/ week of cyanocobalamin will be given , followed by maintenance dose of 15 mcg/ week for rest of 20 weeks.

Anthropometric measurements and dietary information will be collected besides biochemical analysis. IEC sessions will be organized for both the groups.The study hypothesis is that Vitamin B12 supplementation along with iron folic acid (IFA) is more effective in reducing the prevalence of anaemia as compared to IFA supplementation alone.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* Unmarried or married (who still reside with their parents, i.e. prior to 'Gauna') adolescent girl.

Exclusion Criteria:

* Severe anaemia
* Pregnant Adolescent girls
* Medical conditions like TB, Cancer etc

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-11 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin level | at baseline and after 6 months
  The primary outcome would be to assess the change in hemoglobin level after intervention with Iron Folic acid & cyanocobalamin weekly supplementation for 6 months and to compare the results with the group 1 in which only Iron and Folic acid would be supplemented

SECONDARY OUTCOMES:
Change in serum ferritin, folic acid and vitamin B12 levels | at baseline and at end of 6 months
  The secondary outcome would be to assess the change in level of serum ferritin, folic acid and Vitamin B12 after intervention with Iron Folic acid & cyanocobalamin weekly supplementation for 6 months and to compare the results with the group 1 in which only Iron and Folic acid would be supplemented

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gurdayal S Toteja, Ph.D, Principal Investigator — Indian Council of Medical Research; Priyanka Gupta, M.Sc, Principal Investigator — Indian Council of Medical Research; Dr. Neena Bhatia, Ph.D, Principal Investigator — Delhi University; Dr. Naval K Vikram, M.D., Principal Investigator — All India Institute of Medical Sciences; Dr. Anupa Siddhu, Ph.D, Principal Investigator — Delhi University
Locations (1):
- Kirti Nagar Slums, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Basu RN, Sood SK, Ramachandran K, Mathur M, Ramalingaswami V. Etiopathogenesis of nutritional anemia in pregnancy: a therapeutic approach. Am J Clin Nutr. 1973 Jun;26(6):591-4. doi: 10.1093/ajcn/26.6.591. No abstract available. PMID 4575153
- [Background] Sood SK, Ramachandran K, Mathur M, Gupta K, Ramalingaswamy V, Swarnabai C, Ponniah J, Mathan VI, Baker SJ. W.H.O. sponsored collaborative studies on nutritional anaemia in India. 1. The effects of supplemental oral iron administration to pregnant women. Q J Med. 1975 Apr;44(174):241-58. PMID 1103213
- [Background] Gomber S, Agarwal KN, Mahajan C, Agarwal N. Impact of daily versus weekly hematinic supplementation on anemia in pregnant women. Indian Pediatr. 2002 Apr;39(4):339-46. PMID 11976463
- [Background] Kotecha PV, Nirupam S, Karkar PD. Adolescent girls' Anaemia Control Programme, Gujarat, India. Indian J Med Res. 2009 Nov;130(5):584-9. PMID 20090111
- [Background] Agarwal KN, Gomber S, Bisht H, Som M. Anemia prophylaxis in adolescent school girls by weekly or daily iron-folate supplementation. Indian Pediatr. 2003 Apr;40(4):296-301. PMID 12736400
- [Background] Bruner AB, Joffe A, Duggan AK, Casella JF, Brandt J. Randomised study of cognitive effects of iron supplementation in non-anaemic iron-deficient adolescent girls. Lancet. 1996 Oct 12;348(9033):992-6. doi: 10.1016/S0140-6736(96)02341-0. PMID 8855856
- [Background] Ahmed F, Khan MR, Akhtaruzzaman M, Karim R, Marks GC, Banu CP, Nahar B, Williams G. Efficacy of twice-weekly multiple micronutrient supplementation for improving the hemoglobin and micronutrient status of anemic adolescent schoolgirls in Bangladesh. Am J Clin Nutr. 2005 Oct;82(4):829-35. doi: 10.1093/ajcn/82.4.829. PMID 16210713
- [Background] Deshmukh PR, Garg BS, Bharambe MS. Effectiveness of weekly supplementation of iron to control anaemia among adolescent girls of Nashik, Maharashtra, India. J Health Popul Nutr. 2008 Mar;26(1):74-8. PMID 18637530
- [Background] Sen A, Kanani SJ. Impact of iron-folic acid supplementation on cognitive abilities of school girls in Vadodara. Indian Pediatr. 2009 Feb;46(2):137-43. PMID 19242031
- [Background] Shobha S, Sharada D. Efficacy of twice weekly iron supplementation in anemic adolescent girls. Indian Pediatr. 2003 Dec;40(12):1186-90. PMID 14722370
- [Background] Singla PN, Bhardwaj B, Agarwal DK, Agarwal KN. Vitamin B12 and folic acid in preschool anemia. Indian Pediatr. 1985 Jan;22(1):27-33. No abstract available. PMID 4077257
- [Background] Singla PN, Gupta HP, Ahuja C, Agarwal KN. Deficiency anaemias in preschool children--estimation of prevalence based on response to haematinic supplementation. J Trop Pediatr. 1982 Apr;28(2):77-80. doi: 10.1093/tropej/28.2.77. No abstract available. PMID 6763946
- [Background] Mozaffari-Khosravi H, Noori-Shadkam M, Fatehi F, Naghiaee Y. Once weekly low-dose iron supplementation effectively improved iron status in adolescent girls. Biol Trace Elem Res. 2010 Jun;135(1-3):22-30. doi: 10.1007/s12011-009-8480-0. Epub 2009 Aug 4. PMID 19652922
- [Background] Hettiarachchi M, Liyanage C, Wickremasinghe R, Hilmers DC, Abrams SA. The efficacy of micronutrient supplementation in reducing the prevalence of anaemia and deficiencies of zinc and iron among adolescents in Sri Lanka. Eur J Clin Nutr. 2008 Jul;62(7):856-65. doi: 10.1038/sj.ejcn.1602791. Epub 2007 May 16. PMID 17522609
- [Background] Worthington-White DA, Behnke M, Gross S. Premature infants require additional folate and vitamin B-12 to reduce the severity of the anemia of prematurity. Am J Clin Nutr. 1994 Dec;60(6):930-5. doi: 10.1093/ajcn/60.6.930. PMID 7985636